CLINICAL TRIAL: NCT02748850
Title: Evaluation of the Effectiveness of an Aldehyde Inhibitor Dehydrogenases (DIMATE) on the Cell Population Leukemic or Normal Stem
Acronym: DIMATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-42; 2015-A00043-46 (Registry Identifier: ID RCB); RCAPHM15_0066 (Other: APHM)
Record Dates: First submitted 2016-04-13; First posted 2016-04-22 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Leukemia
Keywords: apheresis patients
MeSH Terms: conditions — Leukemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- leukemia patients (Active Comparator): Patients with acute leukemia and / or refractory anemia with excess blasts and comprising a number of blasts in the blood greater than 5% device.
  Interventions: Biological: blood sample
- apheresis patients (Placebo Comparator): patients with non-myeloid hematological malignancy
  Interventions: Biological: Stem cell donation

INTERVENTIONS:
Biological: blood sample — a blood sample 20 milliliter
  Arms: leukemia patients
Biological: Stem cell donation — The volume of stem cells remained in the tube is recovered
  Arms: apheresis patients

SUMMARY:
Aldehyde dehydrogenases (ALDHs) are cellular enzymes responsible for detoxifying aldehyde resulting from the metabolism of endogenous and exogenous xenobiotic cellular constituents. Although ALDHs are considered to play an important role in tumorigenesis, the role of ALDH activity in cancer stem cells, and more particularly that of the acute leukemia must be specified.

Several studies have shown that ALDHs are potent apoptogenic compounds on normal or cancer cells. Therefore, the cells that were damaged and their increased ALDH activity does not die by apoptosis but become highly proliferating. This result is a plausible mechanism for the "evasion of apoptosis", a characteristic shared by many cancer cells.

On this basis, it is proposed an innovative approach to cancer chemotherapy through inhibition of one of the protective mechanisms against apoptosis, ie the increase in ALDH activity than cancer cells put involved in overcoming the lethal effects of damaged roads. ALDHs of inhibitors they may have immediate application as anti -cancer in vivo? The limited experimental data obtained so far on human tumor xenografts in immunodeficient mice and the absence of data on the in vivo toxicology do not allow direct passage to clinical trials. Indeed, some members of the ALDH superfamily are expressed constitutively in some vital organs they protect against the deleterious effects of xenobiotics and adverse endogenous metabolites. Consequently, if ALDHs should be inhibited, of the collateral damages for the normal cells could occur. However, when normal cells have not undergone deleterious exposure, these harmful metabolites are not or in very small quantities, which do not require high levels of ALDH activity, and therefore without harm to the inhibition of cell of these enzymes.

From a hematological point of view, it seems essential to test the therapeutic index of the inhibitor of ALDH DIMATE between normal hematopoietic cells and leukemic stem. Indeed, in the pathophysiology of acute leukemia, the leukemia stem cells are of major importance because they are much more resistant to chemotherapy than more differentiated cells and thus causing the high rate of relapse observed in acute leukemia despite the high rate of complete remission often obtained. In this study, it will be tested in vitro sensitivity of the cluster of differentiation 4 and cluster of differentiation 38 (CD4/CD38) highly purified of leukemic origin or normal to the DIMATE compound. The objective will be to analyze the effects of DIMATE on the parameters of the proliferation, the apoptose, the cytokinins of secretions and the changes transcriptomic in general, in order to better define the therapeutic index of this compound and to determine all the precursory hematopoietic normals and leukaemic cellular effects. The reversible cytostatic of DIMATE effect on normal cells but its irreversible apoptotic effect on cancer cells is an advantage to try to eliminate.

ELIGIBILITY:
Inclusion Criteria:

* Subject, man or woman, whose age is above 18 years
* Subject whose physical and mental condition allows him to understand the information leaflet
* Presenting acute leukemia and / or refractory anemia with excess blasts and blasts with a higher peripheral blood 5%. For leukemic Group
* Subject to benefit from apheresis for autologous stem cell transplantation as part of a non-myeloid hematological malignancy. For the Group Cytapheresis
* Subject affiliated to the social security scheme
* Subject has signed an informed consent
* Subject with a medical examination adapted to the study was conducted

Exclusion Criteria:

* Subject, man or woman, whose age is above 18 years
* Subject previously treated with chemotherapy for his leukemia. For leukemic Group
* Subject considered "vulnerable person" (Major deprived of freedom, under guardianship, pregnant and lactating women and minors)
* Subject refusing to participate in the study
* Subject not having signed an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06-08 (Actual); Primary Completion 2022-06-07 (Estimated); Study Completion 2022-06-07 (Estimated)

PRIMARY OUTCOMES:
Number of cell in apoptose | 48 months
  Cell labeling to differentiate in vitro at least 10-fold (1 log) induction of apoptosis by the DIMATE on stem cells 'normal' (derived from patients who underwent stem cell mobilization for leukapheresis) versus leukemic stem cells taken before any chemotherapy.
Number of cells which shows a rate the ALDH | 48 months
  Normal and leukemic stem cells were incubated with buffer which contains a substrate for ALDH and an efflux inhibitor. The Cells were incubated at 37 ° C for 30 to 60 minutes, which allows the conversion of fluorescence as a function of the cell rate ALDH. They will also be measured by using specific substrates.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No